CLINICAL TRIAL: NCT04837235
Title: Clinical Study of Safety, Tolerability, and Pharmacokinetics of Hemay005 Tablets in Single and Multiple Doses in Healthy Subjects
Brief Title: Multiple Ascending Dose Study to Assess Safety and Pharmacokinetics of Hemay005 In Healthy Subjects
Acronym: Hemay005
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HM005PS1S04
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Hemay005

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 75mg group (Experimental): 15mg/tablet. Five tablets (75mg) each time. Participants will receive a single dose of Hemay005 tablet in Day 1 followed by twice a day of Hemay005 tablet in Day 3~Day8 and single dose in Day9.
  Interventions: Drug: Hemay005
- 90mg group (Experimental): 15mg/tablet. Six tablets (90mg) each time. Participants will receive a single dose of Hemay005 tablet in Day 1 followed by twice a day of Hemay005 tablet in Day 3~Day8 and single dose in Day9.
  Interventions: Drug: Hemay005
- 105mg group (Experimental): 15mg/tablet. Seven tablets (105mg) each time. Participants will receive a single dose of Hemay005 tablet in Day 1 followed by twice a day of Hemay005 tablet in Day 3~Day8 and single dose in Day9.
  Interventions: Drug: Hemay005

INTERVENTIONS:
Drug: Hemay005 — oral

SUMMARY:
Hemay005 is a novel phosphodiesterase type 4(PDE4) inhibitor being developed for the treatment of psoriasis. There were 3 dose cohorts (75mg, 90mg, 105mg) with 12 healthy subjects in each cohorts (6 males and 6 females). This study includes an 11-day Screening Period, a 1-day single dose and 7-days multiple doses Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

1. healthy subjects aged 18 to 60 years, The ratio of male to female is 1:1
2. male Bodyweight（BW）≥ 50kg, female Bodyweight（BW）≥ 45kg, Body mass index (BMI) in 18-28 (including upper and lower limit of the range);
3. All male subjects must agree and commit to the use of a reliable contraceptive regimen(including vasoligation, abstinence, using a condom) for the duration of the study(from screening until 6 months after the last dose), Female participants with a negative pregnancy test (serum) at both the screening visit and at Day-1, Female subjects and female partners of male subjects must agree and commit to the use of a reliable contraceptive regimen ( oral contraceptive medications or non-oral contraceptive medications) for the duration of the study(from screening until 6 months after the last dose);
4. Ability to understand and be willing to sign a written informed consent before study entry;
5. Subjects would have good communication with the investigator and could comply with protocol.

Exclusion Criteria:

1. A history of clinically severe gastrointestinal, hepatic, renal, cardiovascular, dermatological, immunological, respiratory, endocrine, oncological, neurological, metabolic, psychiatric disease or haematological disorders;
2. Have a known history of hypersensitivity to any medicine or food, or allergy to the test article or any of the excipient of the test article;
3. Those who have or are suffering from gastrointestinal, liver and kidney diseases that affect drug absorption or metabolism
4. A history of chronic infection (ie, tuberculosis);
5. A medical history of any clinically significant medical disease or surgery within 4 weeks of the screening
6. Clinically significant laboratory abnormal results at screening or prior to the first dose of study drug;
7. Clinically significant abnormal 12-lead ECG or vital signs
8. Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, hepatitis C virus antibody or Treponema pallidum antibody at screening;
9. Within 1 year before study enrollment of frequent alcohol consumption, defined by average intake of greater than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL of spirits with 40% alcohol content, or 150 mL wine), Participants who are unable to abstain from smoking during the study or quitting smoking for less than 3 months;
10. Positive urine screen for drug and cigarettes, positive breath test for alcohol;
11. Subjects who use soft drugs (ie marijuana )within 3 months of the screening and entire study duration or hard drugs (ie cocaine, phencyclidine ) within 1 year of the screening and entire study duration;
12. Dietary habits or food intolerances which will interfere with the requirements for participants to consume a standardised diet whilst confined to the clinical unit;
13. Participants who eat special food (Including grapefruit and/or Xanthine diet) for 14 days prior to dosing or any caffeine containing food or drinks, i.e. chocolate for 48 hours prior to dosing or drinking alcohol for 24 hours prior to dosing and not will stop to intake above food and drinks;
14. Use of any drug that inhibits or induces hepatic metabolism of drugs within 30 days of planned study drug administration and entire study duration (e.g. inducers: barbiturates, carbamazepine, rifampicin, phenytoin, glucocorticoid and omeprazole; inhibitors-SSRI（Selective serotonin reuptake inhibitors） antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones and antihistamines);
15. Participant who received any medicine within 14 days of the initial dose of study drug;
16. Have received other clinical trials treatment within 3 months prior to study;
17. Participants who have donated of blood (>400 mL) within 4 weeks of the study, or plan to donate of blood during of the study and 4 weeks after the study;
18. Subjects cannot complete the study due to other reasons or by the investigator's judgment;
19. Pregnancy or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs), related AEs and serious AEs (SAEs) | From Day 1 to Day 11
  All subjects who receive the drug will be analyzed for safety, and the safety evaluation will refer to CTCAE 5.0 standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, China